CLINICAL TRIAL: NCT02862704
Title: An Open-label, Uncontrolled, Single-arm Pilot Study to Evaluate Safety and Efficacy of Intratumoral Delivery Mediated MG7-targeted Chimeric Antigen Receptor T Cells in Advanced MG7 Positive Liver Metastases
Brief Title: A Study of MG7 Redirected Autologous T Cells for Advanced MG7 Positive Liver Metastases(MG7-CART)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Shanghai GeneChem Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG7-CART
Record Dates: First submitted 2016-08-07; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Liver Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MG7-CART (Experimental): A single dose of MG7-CART cells will be administered by intra-tumor injection under ultrasound guidance. The dose is 1-6x108 MG7-CAR positive T cells. The infusion will be scheduled to occur 2 days after two doses of 1.5 grams/m2 of cyclophosphamide, which will be administered according to standard procedures. The cells perfusion process would lasts 1min to 2min, and an interventional radiologist would operate the cell infusion.
  Interventions: Biological: MG7-CART

INTERVENTIONS:
Biological: MG7-CART — Ultrasound-guided intra-tumor injection as the route of T cell delivery, so that more T cells gathered at the tumor site, less migrate to the normal tissue, thereby enhancing the efficacy of anti-tumor, reducing the potential of side effects. And MG7-CART is a 2nd CAR, with MG7 as the target protein, 4-1BB as co- stimulator
  Other Names: Ultrasound-guided Intra-tumor Infusion of MG7-CART cells

SUMMARY:
The purpose of this study is to collect the data on the safety and potential effectiveness of intra-tumor injection of MG7-CART cells under ultrasound guidance in patients with liver metastases expressing MG7 positively.

DETAILED DESCRIPTION:
Designer T cells are prepared by PBMC which from patients by leukapheresis, and then activated and re-engineered to express chimeric antigen receptors (CARs) specific for MG7, which is a glycosylated protein of CEA. Cells are expanded in culture and returned to the participant by intra-tumor injection at the dose of (1-6)×108 CAR positive T cells. The cells perfusion process would last for 1min to 2min. The dose of 1.5 grams/m2 of cyclophosphamide will be given two days before CART cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* MG7 expression positive by histologically confirmed;
* Aged between 18 and 69;
* Persistent cancer after at least one prior standard of care chemotherapy, has no willing for surgery or cannot be suitable for surgery patients;
* Tumor is too big to surgical resection;
* Life expectancy greater than 4 months;
* Satisfactory organ and bone marrow function as defined by the following: (1) creatinine <1.5mg/dl; (2) cardiac ejection fraction of >55%; (3) hemoglobin>9g/dl, bilirubin 2.0×the institution normal upper limit;
* Without bleeding disorder or coagulation disorders;
* Dont allergy to Radiocontrast agent;
* Birth control;
* Adequate venous access for apheresis, and no other contraindications for leukapheresis;
* Voluntary informed consent is given.

Exclusion Criteria:

* Pregnant or lactating women;
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary;
* Patients in the situation of: (1) 30 days before apheresis is still in the period of other antitumor drug observation; (2) patient dont recuperate from earlier acute adverse influence brought by any treatments accepted before;
* Four weeks before recruit accepted radiation therapy;
* Previously treatment with any gene therapy products;
* Feasibility assessment during screening demonstrates<30% transduction of target lymphocytes, or insufficient expansion (<5-fold) in response to CD3/CD28 costimulation;
* Any serious, uncontrolled diseases (including, but not limit to, unstable angina pectoris, congestive heart failure, grade III or IV cardiac disease, serious arrhythmia, liver and kidney disorders or metabolic diseases, CNS diseases);
* Patient with severe acute hypersensitive reaction;
* Taking part in other clinical trials;
* Study leader considers not suitable for this tiral.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse event | 6 weeks
  adverse event is evaluated with CTCAE, version 4.0

SECONDARY OUTCOMES:
Number of patients with tumor response | 8 weeks
  summarize tumor response by overal response rates
Detection of transferred T cells in the circulation using quantitative -PCR | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yongzhan Nie, Doctor, Principal Investigator — Xijing Hospital of Digestive Diseases
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided